CLINICAL TRIAL: NCT04568967
Title: Expanding Xpert Ultra Testing for TB Diagnosis Among HIV-positive Patients Admitted to Hospital in Africa
Brief Title: TB-CAPT EXULTANT - HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Instituto Nacional de Saúde, Mozambique (Other Government); Centro de Investigação em Saúde de Manhiça (Other); National Institute for Medical Research, Tanzania (Other Government); Ifakara Health Institute (Other); Ospedale San Raffaele (Other); Swiss Tropical & Public Health Institute (Other); African Society for Laboratory Medicine (Unknown); Heidelberg University (Other); Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TB043-3/1
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Tuberculosis; HIV Coinfection; Diagnoses Disease
MeSH Terms: conditions — Tuberculosis; HIV Infections | interventions — Defecation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): The intervention arm for this trial consists of HIV patients with TB testing performed regardless of presence of TB symptoms. Testing will be done on expectorated sputum, stool and concentrated urine with Ultra, and urine with AlereLAM.
  To fulfil exploratory objectives, we will also collect and store 2x tongue swabs for molecular TB diagnostic assay (Xpert Ultra and/or LumiraDx) testing, blood for testing with CRP, and urine samples which will be stored for retrospective FujiLAM testing and analysis.
  Interventions: Diagnostic Test: Concentrated urine with Xpert Ultra; Diagnostic Test: Stool with Xpert Ultra
- control arm (No Intervention): The control arm for this trial will consist of patients managed according to the current WHO recommended TB testing practices for HIV positive inpatients (as of Q1 2020).
  TB testing will be done as follows:
  Sputum Ultra performed whenever the patient has cough, fever, weight loss over night sweats and/or Ultra performed on any tissue (including lymph nodes) from patients with clinical suspicion of extrapulmonary TB.
  and/or: Urine Alere TB-LAM performed if patients have signs and symptoms of TB (pulmonary and/or extrapulmonary), or with advanced HIV disease, or who are seriously ill, or else irrespective of signs and symptoms of TB, but combined with a CD4 cell count of less than 200 cells/mm .

INTERVENTIONS:
Diagnostic Test: Concentrated urine with Xpert Ultra — Molecular TB diagnostic test on urine
  Arms: intervention arm
Diagnostic Test: Stool with Xpert Ultra — Molecular TB diagnostic test on stool
  Arms: intervention arm

SUMMARY:
The overall aim of this study is to assess the potential of an expanded TB testing strategy to increase the number of HIV-positive patients with microbiologically diagnosed TB who are started on treatment in adult wards of sub-Saharan Africa.

DETAILED DESCRIPTION:
To investigate the effect of an expanded TB screening strategy among HIV-positive patients admitted to hospital (including Ultra on sputum, stool and urine, and AlereLAM on urine, performed regardless of presence of TB symptoms) on the proportion of microbiologically-confirmed TB cases starting treatment within 72 hours of enrolment, compared to Ultra testing (on sputum/any tissue) and AlereLAM (on urine) in only those patients who are symptomatic for TB or fulfilling WHO testing recommendations.

to assess the impact of this screening strategy on 2-month all-cause mortality.

• to assess the feasibility of multiple specimens' collection for TB diagnosis within 72 hours of enrolment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 years old and above)
2. Confirmed HIV infection by serology (including both antiretroviral (ART)- naïve and experienced)
3. Admitted to the hospital (adult medical wards) at the time of enrolment.

Exclusion Criteria:

1. Unable to provide informed consent (if no authorized relatives are in the position to provide the consent)
2. Living outside the catchment area of the participating hospital(s)
3. with plans to migrate outside the catchment area within 2 months after recruitment.
4. Currently receiving anti-TB therapy or having received anti TB therapy in the last 6 months prior to enrolment
5. Receiving preventive TB treatment in the preceding 6 months
6. Patients admitted for traumatic reasons, acute abdomen, delivery (maternal conditions), or for planned/scheduled surgery.
7. Referred from other hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1172 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
proportion of participants diagnosed with microbiologically confirmed TB and started on TB treatment within 72 hours of enrolment | 72 hours after enrolment
  The proportion of participants diagnosed with microbiologically confirmed TB and started on TB treatment within 72 hours of enrolment, separately for intervention and control arm. The numerator is the number of participants per study arm who are diagnosed with microbiologically confirmed TB and start on treatment within 72 hours of enrolment. The denominator is the number of participants enrolled per study arm. We will compare this indicator between both study arms.

SECONDARY OUTCOMES:
Eight-week all-cause mortality | 8 weeks after enrolment
  Eight-week all-cause mortality (main secondary endpoint) among all participants enrolled. The numerator will be number of deaths during eight weeks after enrolment, the denominator is the number of participants enrolled. We will compare this indicator between both study arms.
The proportion of participants who are diagnosed with TB (irrespective of bacteriological confirmation) and started TB treatment within 72 hours of enrolment. | 72 hours after enrolment
  The proportion of participants who are diagnosed with TB (irrespective of bacteriological confirmation) and started TB treatment within 72 hours of enrolment. The numerator is the number of participants diagnosed with TB (with or without bacteriological confirmation) who started treatment within 72 hours of enrolment; the denominator is the number of participants enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto García-Basteiro, MD, Principal Investigator — Barcelona Institute for Global Health
Locations (4):
- Mozambique (2):
  - Centro de Investigação em Saúde de Manhiça-Fundação, Manhiça, Vila Da Manhiça
  - Instituto Nacional de Saúde (INS), Maputo
- Tanzania (2):
  - Ifakara Health Institute (IHI), Bagamoyo
  - National Institute of Medical Research (NIMR), Mbeya

IPD SHARING:
Plan to Share IPD: Yes
Individual, de-identified participant data may be shared, including data dictionaries. Available documents include the study protocol and statistical analysis plan. Templates of the informed consent forms may be shared upon request. The data will be available immediately following publication with no end date, will be shared with anyone who wishes to access them, and will be available for any purpose of analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of the primary peer-reviewed manuscript

REFERENCES:
- [Derived] Mangu C, Cossa M, Ndege R, Khosa C, Leukes V, de la Torre-Perez L, Machiana A, Kivuma B, Mnzava D, Zachariah C, Manjate P, Tagliani E, Schacht C, Buech J, Singh S, Ehrlich J, Riess F, Sanz S, Kranzer K, Cox H, Sabi I, Nguenha D, Meggi B, Weisser M, Ntinginya N, Schumacher S, Ruhwald M, Penn-Nicholson A, Garcia-Basteiro AL; TB-CAPT Consortium. Expanding Xpert MTB/RIF Ultra(R) and LF-LAM testing for diagnosis of tuberculosis among HIV-positive adults admitted to hospitals in Tanzania and Mozambique: a randomized controlled trial (the EXULTANT trial). BMC Infect Dis. 2024 Aug 15;24(1):831. doi: 10.1186/s12879-024-09651-z. PMID 39148008

DOCUMENTS (2):
  • Study Protocol (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT04568967/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT04568967/SAP_001.pdf